CLINICAL TRIAL: NCT05462379
Title: Autologous Heterotopic Fresh Ovarian Graft in Young Woman With Locally Advanced Cervical Cancer Eligible for Pelvic Radiotherapy Treatment
Brief Title: Autologous Heterotopic Fresh Ovarian Graft in Woman With LACC Eligible for Pelvic Radiotherapy Treatment.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MARILIA ALBANEZI BERTOLAZZI (Other)
Responsible Party: Sponsor-Investigator, MARILIA ALBANEZI BERTOLAZZI, Principal investigator/ Gynaecologist, Instituto do Cancer do Estado de São Paulo
Organization: Instituto do Cancer do Estado de São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP1782
Record Dates: First submitted 2022-06-09; First posted 2022-07-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Cervical Carcinoma; Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (No Intervention): 10 patients: Pelvic Chemoradiotherapy
- Ovarian Graft (Experimental): 10 patients: Before the beginning of pelvic radiotherapy, one of the ovaries will be removed by laparoscopy. Ovary slices of 1-2 mm will be prepared in sterile environment and engrafted in the fatty tissue of inner tight. One representative fragment will undergo histologic evaluation. These procedures will be done in the same surgical time.
  Interventions: Procedure: Ovarian graft

INTERVENTIONS:
Procedure: Ovarian graft — Before the beginning of pelvic radiotherapy, one of the ovaries will be removed by laparoscopy. Ovary slices of 1-2 mm will be prepared in sterile environment and engrafted in the fatty tissue of inner tight. One representative fragment will undergo histologic evaluation. These procedures will be done in the same surgical time.
  Other Names: Autologous Heterotopic Fresh Ovarian Graft
  Arms: Ovarian Graft

SUMMARY:
Pelvic chemoradiotherapy (CRT) is an effective treatment for Locally Advanced Cervical Cancer (LACC). However, CRT induces premature ovarian failure ceasing the production of ovarian hormones. This may lead to severe consequences to the patient's life quality, sexuality and overall healthy. An acceptable treatment to minimize the adverse effects caused by the lack of ovarian hormones is hormonal replacement but less than 40% of the patients younger than 50 years have access to this treatment. A second alternative treatment is ovarian transposing which is a surgical technique with variable success rate depending on how far the ovaries are from the radiotherapy field. A third, more promising, alternative is involves using autologous ovarian tissue as a graft in tissues far from the radiotherapy field. This treatment has the potential of maintaining the natural ovarian hormones production at a lower-cost and requiring a simpler procedure. The primary objective of this randomized phase 1-2 clinical trial is to validate the feasibility of ovarian tissue engraft into fatty tissue and its endocrine functionality.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of squamous cell carcinoma or adenocarcinoma of the cervix.
* FIGO 2018 staging IB3 to IVA.
* Absence of ovarian involvement.
* Age ≤35 Years.
* Absence of metastatic disease.
* Written consent.

Exclusion Criteria:

* Previous treatment for cervical cancer or other malignant diseases.
* Rare histology tumors.
* Absence of one or both ovaries.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Dosage of serum levels of follicle stimulating hormone (FSH) in mUI/ml in intervention (engraft of ovarian tissue into fatty tissue) and control groups. Dosage will be performed at baseline and post radiotherapy (2, 6, 12 and 24 months). | 2 years
  Endocrine functionality is defined as FSH levels under 25 mUI/ml.
Dosage of serum levels of estradiol in pg/ml in intervention (engraft of ovarian tissue into fatty tissue) and control groups. . Dosage will be performed at baseline and post radiotherapy (2, 6, 12 and 24 months). | 2 years
  Endocrine functionality is defined as estradiol upper 47 pg/mL.

SECONDARY OUTCOMES:
Dosage of serum levels of glucose in mg/dL in intervention and control groups. (Time frame: At baseline and post radiotherapy month 2, 6, 12 and 24). | 2 years
  Evaluation of glucose metabolism.
Measure of serum glycated hemoglobin in percentage in intervention and control groups. (Time frame: At baseline and post radiotherapy month 2, 6, 12 and 24). | 2 years
  Evaluation of glucose metabolism.
Measure of serum levels of cholesterol in mg/dL in intervention and control groups. (Time frame: At baseline and post radiotherapy month 2, 6, 12 and 24). | 2 years
  Evaluation of lipid metabolism.
Measure of serum levels of triglycerides in mg/dL in intervention and control groups. (Time frame: At baseline and post radiotherapy month 2, 6, 12 and 24). | 2 years
  Evaluation of lipid metabolism.
Evaluate the changes in bone mineral density (BMD) in femoral neck and lumbar spine by bone densitometry, evaluating T and Z scores standard deviation (SD) in intervention and control groups. Time frame: At baseline and post radiotherapy month 12 and 24. | 2 years
Bioimpedance monitoring to evaluate changes in body composition by fat and lean mass percentage in intervention and control groups. Time frame: At baseline and post radiotherapy month 12 and 24). | 2 years
Quantification of body mass index reported in kg/m2 in intervention and control groups. Time frame: At baseline and post radiotherapy month 12 and 24). | 2 years
  Evaluation of changes in body mass.
Score life quality in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ C30) in intervention and control groups. | 2 years
  EORTC QLQ C30 was developed and validated to assess the quality of life of cancer patients.
  The 30-item EORTC QLQ-C30 is a disease-specific measure that assesses multiple QoL domains in patients with cancer. There are five functioning scales that measure physical, role, emotional, cognitive, and social functioning. Three symptom scales measure fatigue, pain, and nausea/vomiting.
Score life quality in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 Cervical Cancer Module (EORTC QLQ C30 CX24) in intervention and control groups. | 2 years
  EORTC QLQ-CX24 Scoring Manual The Cervical Cancer Module is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. The EORTC QLQ-CX24 was designed to assess disease-specific and treatment-specific aspects of QoL in patients with cervical cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Cancer do Estado de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

DOCUMENTS (1):
  • Informed Consent Form (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT05462379/ICF_001.pdf